CLINICAL TRIAL: NCT00669760
Title: Dissection of Staphylococcus Aureus Infection From Colonization in Cystic Fibrosis Patients, a Non-interventional, Prospective, Longitudinal Multicenter Study.
Brief Title: Dissection of Staphylococcus Aureus Infection From Colonization in Cystic Fibrosis Patients
Acronym: StaphCI
Status: Completed | Type: Observational
Sponsor: University Hospital Muenster (Other)
Collaborators: Mukoviszidose eV Bonn Germany (Unknown)
Responsible Party: Principal Investigator, Barbara Kahl, Prof. Dr. Barbara Kahl, University Hospital Muenster
Other Study IDs: Muko e.V. S05/07
Record Dates: First submitted 2008-04-28; First posted 2008-04-30 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2015-01

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; Staphylococcus aureus; persistent colonization-infection; clinical status; lung function
MeSH Terms: conditions — Cystic Fibrosis; Staphylococcal Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — Sera
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: CF-patients with persistent culture of Staphylococcus aureus in their respiratory specimens
  Interventions: Other: non-interventional study

INTERVENTIONS:
Other: non-interventional study — does not apply
  Other Names: does not apply

SUMMARY:
Staphylococcus aureus is not only one of the first pathogens infecting the airways of cystic fibrosis (CF) patients, but also a highly prevalent microorganism (>60% of all CF patients; European and American CF registries; (4,25), which often persists for several years in the respiratory tract of CF patients.

The purpose of this study is to dissect infection by S. aureus from colonization. Therefore, the following non-interventional prospective, longitudinal multicenter study will be conducted to develop the following hypothesis:

CF patients with high bacterial loads are more likely to be infected by S. aureus than patients with low bacterial loads.

Primary endpoint: bacterial load of sputum cultures

Secondary endpoints:

* nasal carriage
* molecular analysis of S. aureus (Monoclonal/polyclonal)
* serum: S. aureus-specific antibodies, S100A12, IL-8, TNF-alpha
* sputum: S100A12, IL-8, myeloperoxidase
* S. aureus therapy regimens
* lung function tests: FEV1, deltaFVC , deltaMEF25
* BMI development

Inclusion criteria: S. aureus cultures for more than 6 months within the last year, children (>6 years) and patients, who are able to perform lung function tests Exclusion criteria: P. aeruginosa and/or B. cepacia cultures from the specimens for more than 6 months within the last year before recruitment or during the study period In addition to microbiological investigations and clinical laboratory tests, the actual clinical situation will be evaluated and reported during the study period. The results of this observational study will be used to carefully plan a clinical interventional study. Furthermore, with the results it might be possible to characterize a subpopulation of patients, which is at greater risk for S. aureus infections.

DETAILED DESCRIPTION:
Protocol synopsis Title: Dissection of Staphylococcus aureus infection from colonization in cystic fibrosis patients. A non-interventional prospective, 2-year longitudinal multicenter study

Study objectives: The aim of the study is to dissect S. aureus infection from colonization of the pathogen in airway secretions of CF patients during a 2 year period by means of a non-interventional, prospective, longitudinal multicenter study.

The following hypothesis will be developed:

CF patients with high bacterial loads are more likely to be infected by S. aureus than patients with low bacterial loads.

Definition of infection:

* change in volume, colour or consistency of sputum (exacerbation)
* increased cough
* malaise, fatigue or lethargy
* body temperature more than 38°C
* new or increased hemoptysis
* anorexia or weight loss
* sinus pain or tenderness
* change in sinus discharge
* change in chest sounds
* ten percent decrease in pulmonary function from a previous recorded value (FEV1, MEF25)
* radiographic changes indicative of pulmonary infection

Primary endpoint: bacterial load of sputum cultures [high (>/= 106CFU/ml); low (<106CFU/ml)]

Secondary endpoints are:

* assessment of nasal S. aureus carriage
* serum samples: antibody titres against S. aureus specific antigens; S100A12, IL-8,TNF-alpha, CRP
* molecular analysis of S. aureus colonization/infection (monoclonal or heteroclonal)
* sputa analysis: activity of S100A12, IL-8 and myeloperoxidase
* antibiotic treatment regimens against S. aureus
* body mass index
* lung function tests: FEV1, deltaFVC, deltaMEF25

Extensive microbiological investigations will be performed when the patients are seen at their regular visits in the outpatient clinics or if exacerbations occur. During the study period of 2 years, at least 8 visits to the outpatient clinic should be recorded. The following clinical parameters will be documented:

* lung function
* body mass index (weight/height)
* antibiotic treatment Diagnosis: CF and positive S. aureus cultures for more than 6 months within the last year Localisation of the study: multicenter study in Germany Number of centers: Seven centres agreed already to participate in the study. More centers have been and will be contacted.

Design: non-interventional prospective, longitudinal multicenter study Planned number of patients/volunteers: 228 Inclusion criteria: positive S. aureus cultures for more than 6 months within the last year; children (>6 years) and patients with CF, who are able to perform lung function tests Exclusion criteria: Pseudomonas aeruginosa and/or Burkholderia cepacia colonization or infection for more than 6 months within the last year before recruitment; patients who have not been colonized with these pathogens before but acquire them within the study period and are colonized/infected for more than 6 months during the observation period

ELIGIBILITY:
Inclusion Criteria:

* positive S. aureus cultures for more than 6 months within the last year; children (>6 years) and patients with CF, who are able to perform lung function tests

Exclusion Criteria:

* Pseudomonas aeruginosa and/or Burkholderia cepacia colonization or infection for more than 6 months within the last year before recruitment; patients who have not been colonized with these pathogens before but acquire them within the study period and are colonized/infected for more than 6 months during the observation period

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: CF-patients with persistent S. aureus culture in their airway specimens
Sampling Method: Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2008-07; Primary Completion 2011-07 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
bacterial load of sputum cultures [high (>/= 1000000CFU/ml); low (<1000000CFU/ml)] | 2 years

SECONDARY OUTCOMES:
antibody titres against S. aureus specific antigens; S100A12, IL-8, TNF-alpha, CRP | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Barbara C Kahl, MD, Principal Investigator — Dept. Med. Microbiology, University Clinics Muenster, Germany
Locations (17):
- Medizinische Universität Innsbruck, Innsbruck, Austria
- Germany (16):
  - Charite Berlin Campus Benjamin Franklin, Berlin
  - Clinic for Children and Adolescents Ruhr University Bochum St Josef Hospital, Bochum
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Heinrich-Heine University Duesseldorf, Düsseldorf
  - University Clinics Essen, Essen
  - Ruhrlandklinik Essen-Heidhausen, Essen
  - Universitätsklinikum Halle, Halle
  - Dres Heuer-Runge-Sextro, Hamburg
  - Medical School Hannover, Hanover
  - University Clinics Jena, Jena
  - Children's Hospital Park Schoenfeld, Kassel
  - Universitätsklinikum Leipzig, Leipzig
  - University Clinics Muenster, Münster
  - Clemenshospital, Münster
  - Children's Hospital Osnabrueck, Osnabrück
  - University Clinics Tuebingen, Tübingen

REFERENCES:
- [Derived] Junge S, Gorlich D, den Reijer M, Wiedemann B, Tummler B, Ellemunter H, Dubbers A, Kuster P, Ballmann M, Koerner-Rettberg C, Grosse-Onnebrink J, Heuer E, Sextro W, Mainz JG, Hammermann J, Riethmuller J, Graepler-Mainka U, Staab D, Wollschlager B, Szczepanski R, Schuster A, Tegtmeyer FK, Sutharsan S, Wald A, Nofer JR, van Wamel W, Becker K, Peters G, Kahl BC. Factors Associated with Worse Lung Function in Cystic Fibrosis Patients with Persistent Staphylococcus aureus. PLoS One. 2016 Nov 18;11(11):e0166220. doi: 10.1371/journal.pone.0166220. eCollection 2016. PMID 27861524